CLINICAL TRIAL: NCT04538287
Title: AtaCor Subcostal Temporary Extravascular Pacing III Study
Acronym: STEP III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DOC-10092
Record Dates: First submitted 2020-08-25; First posted 2020-09-04 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Conduction Defect
Keywords: Temporary Ventricular Pacing
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- AtaCor StealthTrac Lead Model AC-1010 (Active Comparator): Subjects inserted with the AtaCor StealthTrac Lead Model AC-1010. This was the first model evaluated in the study.
  Interventions: Device: AtaCor StealthTrac Lead
- AtaCor StealthTrac Lead Model AC-1020 (Active Comparator): Subjects inserted with the AtaCor StealthTrac Lead Model AC-1020. This was the second model evaluated in the study.
  Interventions: Device: AtaCor StealthTrac Lead
- AtaCor StealthTrac Lead Model AC-1021 (Active Comparator): Subjects inserted with the AtaCor StealthTrac Lead Model AC-1021. This was the third model evaluated in the study.
  Interventions: Device: AtaCor StealthTrac Lead
- AtaCor StealthTrac Lead Model AC-1012 (Active Comparator): Subjects inserted with the AtaCor StealthTrac Lead Model AC-1012. This is the fourth model currently being evaluated in the study.
  Interventions: Device: AtaCor StealthTrac Lead

INTERVENTIONS:
Device: AtaCor StealthTrac Lead — Subjects are assigned non-randomly to receive one of the four AtaCor StealthTrac leads being evaluated in the study.

SUMMARY:
Third in-human study for the AtaCor Extravascular (EV) Temporary Pacing Lead System to collect initial safety and performance data for the latest AtaCor System.

The objective of the study is to generate safety and performance data of the latest AtaCor EV Temporary Pacing Lead System 1) to support the development a future pivotal study with an indication limited to a maximum of 7 days, and 2) to obtain early clinical data for future research related to longer-term use.

DETAILED DESCRIPTION:
Prior revisions of the study intended to evaluate multiple StealthTrac Leads (Models AC-1010, AC-1020, AC-2021 and AC-1030) to support the development of a future pivotal study. In the most recent revision of the study, an additional StealthTrac Lead (Model AC-1012) will be evaluated to support use in a larger pivotal study.

This study is a feasibility study serving dual purposes: 1) to generate developmental clinical data in support of a subsequent pivotal clinical study and marketing application for temporary pacing (in patients that retain the lead for a maximum of 7 days); and 2) to obtain early data for future research related to longer-term use (in patients that retain the lead for a maximum of 14 days).

Subjects undergoing a qualifying index procedure will have a Model AC-1012 StealthTrac Lead inserted, evaluated for a Maximum Lead Insertion Time prior to removal and a final post-removal follow-up 27-33 days after lead insertion. The following elements will change after the absence of AtaCor-related cardiac tamponade and no more than one (1) serious AtaCor-related pericardial effusion has been confirmed from the initial eight (8) experiences with the Model AC-1012 StealthTrac Lead, including insertion and removal procedures performed by multiple operators:

* Maximum Lead Insertion Time will change from 7 to 14 Days
* Follow-up will change from in-hospital follow-up only to allowing hospital discharge with the StealthTrac lead inserted, but capped and inactive after Day 2 provided in-person wound checks occur at least every 3 days
* Echocardiography requirements will transition from 3 distinct days to procedure day and removal day only.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Indicated for closed-chest cardiac invasive procedure (e.g. transcatheter valve replacement, balloon valvuloplasty, permanent pacemaker implantation and pacing lead extractions/revisions)

Exclusion Criteria:

1. NYHA IV functional class
2. Oxygen dependency
3. BMI ≥ 35 kg/m2
4. Circumstances that prevent data collection or follow-up (e.g., inability to perform a short walk with the Holter monitor)
5. Participation in any concurrent clinical study without prior written approval from the Sponsor
6. Inability to give an informed consent to participate in the Study

   Known prior history for any of the following:
7. Median or partial sternotomy
8. Surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium
9. Significant anatomic derangement of or within the thorax (e.g., pectus excavatum, significant scoliosis)
10. Thoracic radiation therapy, pneumothorax, pneumomediastinum or other medical treatments/conditions which may complicate the AtaCor EV Temporary Pacing Lead System insertion procedure
11. Pericardial disease, pericarditis and mediastinitis
12. Medical treatments, surgeries or conditions that increase the potential for pericardial adhesions
13. Severe to very severe airflow limitation, defined as FEV1/FVC <0.7 AND FEV1 < 50% predicted
14. Symptomatic COPD exacerbation associated with either:

    1. Modified MRC Dyspnea Scale Grade ≥2, OR
    2. CAT Assessment
15. Surgically corrected congenital heart disease (not including catheter-based procedures)
16. Allergies to the device materials such as stainless steel, titanium, platinum, iridium, polyethylene, polyurethane, polycarbonate and silicone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-10-03 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Safety - Freedom from Adverse Device Effects | Lead removal (up to 14 Days)
  Freedom from Adverse Device Effects (ADE)
Performance - Pacing Capture Threshold | Lead removal (up to 14 Days)
  Summary statistics for pacing capture threshold for each StealthTrac Lead model from insertion through removal
Performance - Pacing Impedance | Lead removal (up to 14 Days)
  Summary statistics for pacing impedance for each StealthTrac Lead model from insertion through removal for each StealthTrac Lead model from insertion through removal
Performance - Sensed R-wave Amplitude | Lead removal (up to 14 Days)
  Summary statistics for sensed R-wave amplitude for each StealthTrac Lead model from insertion through removal

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Burke, DO, Principal Investigator — AtaCor Medical, Inc.
Locations (4):
- Na Homolce Hospital, Prague, Czechia
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Wellington Regional Hospital, Wellington
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No